CLINICAL TRIAL: NCT00260260
Title: The Pharmacogenetics of Oxycodone Analgesia in Postoperative Pain
Brief Title: OXY-1: The Pharmacogenetics of Oxycodone Analgesia in Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2005-001145-42
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone

INTERVENTIONS:
Drug: Oxycodone

SUMMARY:
Patients undergoing surgery (thyroidectomy and hysterectomy) will postoperatively receive oxycodone intravenously (IV) as pain management with morphine as an escape medicine, if there is insufficient pain relief with oxycodone. Patients' pain and side effects will be registered and after 24 hours they will answer a questionnaire. All included patients will be genotyped accordingly to CYP2D6 and relevant single nucleotide polymorphisms (SNPs), and measures of plasma levels of oxycodone will be performed.

DETAILED DESCRIPTION:
Oxycodone is a semi-synthetic opioid with an analgesic effect in the postoperative pain management comparable to morphine. Oxycodone is N-demethylated by CYP2D6 to its active metabolite oxymorphone, a potent μ-receptor agonist. A genetic polymorphism divides a Caucasian population into two groups: 8% with an enzyme lacking activity, poor metabolizers (PM) and the rest with normal CYP2D6 activity, extensive metabolizers (EM).

Many different, single nucleotide polymorphisms (SNPs) are responsible for interindividual differences in the effect of opioids. Among these are the A118G SNP in the μ-receptor gene OPRM1 and the C3435T and G2677T/A SNPs in the MDR-1 gene of P-glycoprotein. P-glycoprotein is responsible for the absorption, excretion and transport of many drugs including opioids over the blood-brain barrier.

The patients will receive the first Oxycodone dosis of 5 mg iv at the end of the surgery. If their pain is not sufficiently relieved they can be given maximum two times Oxycodone 5 mg iv in the recovery room. If still not sufficiently pain relieved they will be given escape medication (Morphine 5 mg iv) until sufficient pain relief.

Further pain treatment will be by Patient Controlled Analgesia (PCA) with bolus doses of Oxycodone 2 mg iv.

During the first 24 hours postoperatively the patients pain and side effects will be registered.

Three blood samples will be drawn: 1. approximately 30 minutes after first Oxycodone dosis, 2. before leaving the recovery room a couple of hours after surgery and 3. 24 hours after surgery. From these samples plasma levels of Oxycodone and its metabolites will be determined and the genotype of CYP2D6 and the above mentioned SNPs will be determined.

The patients will be divided into two groups: Responder and Non-responder. The Responders are characterized by no use of escape medication (morphine) and satisfaction with pain management in final questionnaire. The Non-responders are characterized by use of escape medicine and/or dissatisfaction with pain management in final questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80 years old
* Caucasian race
* Signed informed consent
* Patients admitted for one of the following operations: thyroidectomy, mastectomy, hysterectomy, mammaexpander operation, nasal septum correction and jaw operations.

Exclusion Criteria:

* Allergy towards oxycodone
* Previous daily opioid use
* Known severe illness (terminal cancer, severe dementia, uncompensated heart failure, kidney failure, liver failure and severe lung failure)
* Lack of ability to use patient controlled analgesia or to follow the trial protocol
* Pregnancy
* Severe psychiatric illness
* Alcoholism
* Ongoing treatment with potent CYP2D6 inhibitors (fluoxetine, paroxetine and terbinafine)
* Severe perioperative complications or re-operation within the first 24 hours
* Use of extra pain management during the anaesthesia with an effect after the operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Responder (satisfaction with pain treatment in questionnaire and no escape medication)
Non-responder (dissatisfaction with pain management in questionnaire and/or escape medication)
Responder status compared to CYP2D6 genotype

SECONDARY OUTCOMES:
Registration of pain, side effects and total amount of oxycodone given compared to CYP2D6 genotype and SNPs

CONTACTS AND LOCATIONS:
Overall Officials: Stine T. Zwisler, Dr., Principal Investigator — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense C, Odense, Denmark